CLINICAL TRIAL: NCT03494101
Title: Interaction Between Non-typhoid Salmonella, Host Microbiota, and Immune System During Acute Infection and Remission
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: SALMONELLA Study
Record Dates: First submitted 2018-03-01; First posted 2018-04-11 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Salmonella Infection Non-Typhoid
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-typhoid Salmonella infection: Patients with a non-typhoid Salmonella infection. Blood samples, stool samples and clinical information will be collected.
  Interventions: Other: Blood samples; Other: Stool samples; Other: Clinical information
- Acute, infectious diarrhea: Patients with acute, infectious diarrhea without non-typhoid Salmonella infection. Blood samples, stool samples and clinical information will be collected.
  Interventions: Other: Blood samples; Other: Stool samples; Other: Clinical information
- Healthy individuals: Healthy individuals with no symptoms of acute or chronic diarrhea. Blood samples, stool samples and clinical information will be collected.
  Interventions: Other: Blood samples; Other: Stool samples; Other: Clinical information

INTERVENTIONS:
Other: Blood samples — Blood samples will be collected and analyzed at different study time points
Other: Stool samples — Stool samples will be collected and analyzed at different study time points
Other: Clinical information — Clinical information will be collected at different study time points using questionnaires

SUMMARY:
Stool and blood samples from patients with a non-typhoid Salmonella infection will be collected during an observation period of six months and analyzed for changes in the microbiota diversity and composition, mutation rates in the Salmonella strains and the specific immune response evoked by the infection. Findings are compared to healthy individuals and individuals with acute, infectious diarrhea caused by other microorganisms.

DETAILED DESCRIPTION:
Infection processes of a non-typhoid Salmonella infection in humans are not well understood and so far, only little research has been conducted in this area. Findings from preclinical studies, using mouse models, attributed a fundamental role in infection control to the gut microbiota and the host immune system (antibody response). In mouse models a non-typhoid Salmonella infection provokes a pronounced antibody response and salmonella-inflicted gut inflammation alters the microbiota diversity and composition in the gut lumen. To date there is only scarce evidence on similar effects in humans.

During the study, longitudinal stool and blood samples will be collected from patients with a non-typhoid Salmonella infection at different study time points (2 weeks, 4 weeks and 6 months after positive Salmonella stool culture) and analyzed for changes in the microbiota, mutation rates in the Salmonella strains and the specific immune response evoked by the infection (e.g. anti-bodies). At each study time point clinical information will be investigated with a questionnaire to assess current symptoms, medication etc. Findings will be compared to healthy individuals and patients with acute, infectious diarrhea caused by other microorganisms than non-typhoid Salmonella.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria:

* Signed informed consent.
* Ability to understand and follow study procedures and understand informed consent
* Age 18-75 years.

Inclusion criteria for patients with non-typhoid Salmonella infection (n=20)

* Acute diarrhea (≥3 bowel movements per day for ≤4 weeks)
* Stool cultures positive for non-typhoid Salmonella ≤4 weeks before inclusion

Inclusion criteria for patients with acute, infectious diarrhea without non-typhoid Salmonella infection (n=10)

* Acute diarrhea (≥3 bowel movements per day for ≤4 weeks)
* Stool cultures negative for non-typhoid Salmonella infection within ≤ 4 weeks

Inclusion criteria for healthy volunteers (n=10)

• No symptoms of acute or chronic diarrhea (2 bowel movements per week to 2 per day)

Exclusion Criteria:

* Current use of antibiotics
* Medication with immunosuppressants (e.g. corticoids, biological therapy).
* Major medical/surgical/psychiatric condition requiring ongoing management. Minor well controlled conditions (i.e. medically controlled arterial hypertension, occupational asthma) may be present.
* Major diagnosis known to chronically affect gut microbiota (e.g. inflammatory bowel disease, liver cirrhosis, colon carcinoma, systemic sclerosis).
* Current diagnosis of a hematological disorder (e.g. severe anemia with hemoglobin <7 g/dl, leukemia) or any other absolute contraindication for blood donation.
* Participation in other clinical study interfering with study procedures.
* Inability to understand study procedures in order to provide inform consent.
* Previous participation in the same study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 patients with a non-typhoid Salmonella infection, 10 patients with acute, infectious diarrhea without non-typhoid Salmonella infection, 10 healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Genomic mutations in non-typhoid Salmonella strains | 4 weeks after index stool culture
  Analyze the evolution of non-typhoid Salmonella during acute infection and remission in humans. The primary variable of interest is the number of observed genomic mutations in non-typhoid Salmonella strains.

SECONDARY OUTCOMES:
Quantification of non-typhoid Salmonella genes associated with: tissue invasion, antibiotic resistance and virulence factors | 4 weeks after index stool culture
  Total number of Salmonella genes associated with tissue invasion Total number of antibiotic resistance genes Total number of virulence factor genes
Identification of most frequently mutated surface antigenes of non-typhoid Salmonella | 4 weeks after index stool culture
  Identification of escape mechanisms of non-typhoid Salmonella (i.e. mutation of surface antigens) to avoid specific immune responses (i.e. antibodies) during acute infection and remission.
Gen Cluster Expression | 2 weeks, 4 weeks and 6 months after index stool culture
  Identification of Salmonella gene clusters expressed during early phases of infection compared to remission.
Mutated non-typhoid Salmonella strains | 4 weeks and 6 months after index stool culture
  Quantification of mutated non-typhoid Salmonella strains that escape specific immune responses.
Microbiota changes | 2 weeks, 4 weeks and 6 months after index stool culture
  Composition (i.e. number of bacteria species identified) and relative diversity of the gut microbial community during acute non-typhoid Salmonella infection and remission. Findings will be compared to changes occurring in the microbiota of healthy individuals and individuals with acute, infectious diarrhea caused by microorganisms other than Salmonella.
Antibody producing cells | 2 weeks and 4 weeks after index stool culture
  Composition (i.e. number of antibody-producing cells) and relative diversity of antibody-producing cells specific for non-typhoid Salmonella.
Antibody producing B-cell clones | 4 weeks after index stool culture
  Number of antibody-producing cell clones (and their corresponding antibodies) against non-typhoid Salmonella isolated from peripheral blood B cells of subjects during remission. Measured variable: Number of Salmonella-specific B-cells per ml blood 4 weeks after infection.
Antibody repertoire | 2 weeks and 4 weeks after index stool culture
  Identification of the antibody repertoire against non-typhoid Salmonella during acute infection in peripheral blood. Measured variable: Antibody titers against various non-typhoid Salmonella strains.
Antigen- Antibody recognition | 4 weeks and 6 months after index stool culture
  Number of antigens of non-typhoid Salmonella recognized by the antibodies isolated from the previous endpoint.
Development of irritable bowel syndrome | End of observational period (6 months)
  Number of patients who develop an irritable bowel syndrome after a non-typhoid Salmonella infection.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Misselwitz, PD Dr.med., Principal Investigator — Division of Gastroenterology, University Hospital Zurich Zurich, Switzerland, 8091
Locations (1):
- Division of Gastroenterology, University Hospital Zurich, Zurich, Switzerland